CLINICAL TRIAL: NCT03504020
Title: ECG Belt for CRT Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECG Belt for CRT Response
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ECG Belt (Experimental): The ECG Belt arm will utilize the ECG Belt Research System at implant and all follow up visits.
  Interventions: Device: ECG Belt Research System
- Control Arm (No Intervention): Standard CRT through 6 months follow-up.

INTERVENTIONS:
Device: ECG Belt Research System — The ECG Belt Research System is used to identify the best vector and programming parameters.
  Arms: ECG Belt

SUMMARY:
The purpose of this clinical study is to compare ECG Belt Research System managed cardiac resynchronization therapy (CRT) patients and a control CRT group with respect to left ventricular (LV) remodeling.

DETAILED DESCRIPTION:
The ECG Belt study is a prospective, interventional, randomized, multi-center, investigational, pre-market research study. The ECG Belt Research System will be used at implant and follow-up to help implanters choose a suitable LV pacing site within the recommended locations for LV lead implantation and optimize pacing vector/timing parameters.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for CRT, with QRS duration ≥130 ms, and planned to be implanted with a market-released Medtronic CRT device with AdaptivCRT and a Medtronic quadripolar LV lead.
* Meets at least one of the following criteria: QRS duration < 150 ms, Prior documented Myocardial Infarction, Non-LBBB
* LVEDD ≥ 55 mm, as determined by site

Exclusion Criteria:

* Permanent/persistent AF or presenting with AF
* Pre-existing or previous LV lead or other confounding devices e.g. Left Ventricular Assist Device, Vagal Nerve Stimulator
* Currently implanted with IPG or ICD with > 10% RV pacing
* Permanent complete AV block
* Enrolled in a concurrent study that may confound the results of this study. Pre-approval from the study manager is required for enrollment of a patient that is in a concurrent study.
* Less than 1 year life expectancy
* Vulnerable adults
* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ECG Belt for CRT Response Clinical Research Specialist, Study Chair — Medtronic
Locations (43):
- United States (34):
  - Hartford Hospital, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Florida Hospital Cardiovascular Research Institute, Orlando, Florida
  - BayCare Health System, Tampa, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - Heartland Cardiology, Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Atrium Health's Carolina Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Mount Carmel East, Columbus, Ohio
  - OhioHealth Research and Innovation Institute (OHRI), Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital- Cedar Crest, Allentown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Vanderbilt University medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Health Research & Education Institute, Fort Worth, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Aurora St. Lukes, Milwaukee, Wisconsin
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis-campus aalst, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- Italy (2):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Istituto Auxologico Italiano - Istituto Scientifico Ospedale San Luca, Milan
- Maastricht Universitair Medisch Centrum (MUMC), Maastricht, Netherlands
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rickard J, Jackson K, Biffi M, Vernooy K, Bank A, Cerkvenik J, Ghosh S, Gold MR. The ECG Belt for CRT response trial: Design and clinical protocol. Pacing Clin Electrophysiol. 2020 Oct;43(10):1063-1071. doi: 10.1111/pace.13985. Epub 2020 Sep 1. PMID 32537740
- [Result] Rickard J, Jackson K, Gold M, Biffi M, Ziacchi M, Silverstein J, Ramza B, Metzl M, Grubman E, Abben R, Varma N, Tabbal G, Jensen C, Wouters G, Ghosh S, Vernooy K; ECG Belt for CRT Response Study Group. Electrocardiogram Belt guidance for left ventricular lead placement and biventricular pacing optimization. Heart Rhythm. 2023 Apr;20(4):537-544. doi: 10.1016/j.hrthm.2022.11.015. Epub 2022 Nov 25. PMID 36442824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * 498 pts enrolled, 55 exits prior to randomization
  * 443 pts randomized, 35 pts not implanted
Groups:
- ECG Belt: The ECG Belt arm will utilize the ECG Belt Research System at implant and all follow up visits.
  >
  > ECG Belt Research System: The ECG Belt Research System is used to identify the best vector and programming parameters.
Period: Overall Study
Arm/Group | ECG Belt | Control Arm
Started | 200 | 208
Completed | 161 | 172
Not Completed | 39 | 36

BASELINE CHARACTERISTICS:
Groups:
- ECG Belt: The ECG Belt arm will utilize the ECG Belt Research System at implant and all follow up visits.>
  > ECG Belt Research System: The ECG Belt Research System is used to identify the best vector and programming parameters.
- Total: Total of all reporting groups
Arm/Group | ECG Belt | Control Arm | Total
Number analyzed (Participants) | 200 | 208 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.4) | 67.8 (10.1) | 68.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 156 | 167 | 323
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End Systolic Volume (LVESV) From Baseline to 6 Months Post-implant.
Description: Relative (%) change in LVESV from the baseline measurement to the 6 month measurement.
Time Frame: baseline to 6 months
Population: Patients were only included in the analysis if they completed the Baseline and 6-month visit. For some patients, if the 6-month visit was not available, but the 9-month visit was, then the 9-month visit was used.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | ECG Belt | Control Arm
Number analyzed (Participants) | 163 | 175
Percent Change | -11.7 (29.0) | -14.7 (29.6)

ADVERSE EVENTS:
Time Frame: Enrollment- 9 months
Groups:
- Control Arm: Standard CRT through 9 months follow-up.
Arm/Group | ECG Belt | Control Arm
All-Cause Mortality (participants affected / at risk) | 12/200 | 6/208
Serious Adverse Events (participants affected / at risk) | 68/200 | 52/208
Other Adverse Events (participants affected / at risk) | 0/200 | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECG Belt (N=200) | Control Arm (N=208)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Accelerated Idioventricular Rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Acute Left Ventricular Failure (Cardiac disorders) | 2 (4) | 5 (5)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmic Storm (Cardiac disorders) | 3 (3) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 3 (3)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac Failure (Cardiac disorders) | 10 (11) | 7 (17)
Cardiac Failure Acute (Cardiac disorders) | 9 (10) | 2 (3)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 8 (10) | 4 (4)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 2 (3) | 1 (1)
Chronic Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 2 (3) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 5 (6) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 2 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 1 (1)
Unevaluable Event (General disorders) | 0 (0) | 1 (1)
Transplant Rejection (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis Enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Infection (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2)
Pneumonia Escherichia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 2 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cauda Equina Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Device Lead Damage (Product Issues) | 1 (1) | 0 (0)
Lead Dislodgement (Product Issues) | 4 (4) | 6 (6)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 1 (1)
End Stage Renal Disease (Renal and urinary disorders) | 2 (3) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (2) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site will not independently publish, publicly disclose, present or discuss any results of or information pertaining to the study until a multi-center publication is released; provide however that if a multi-center publication is not released within 1 year after completion of the study at all sites involved in the study, Study Site will have the right to publish the results of, and information pertaining to , their activities conducted under their CTA, in accordance with provision of CTA.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT03504020/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03504020/SAP_002.pdf